CLINICAL TRIAL: NCT02724943
Title: Systems Approach to Obesity Prevention in Underserved Children in Texas (Randomized Controlled Trial)
Brief Title: Texas Childhood Obesity Research Demonstration (TX CORD) Project
Acronym: TXCORDRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Baylor College of Medicine (Other); Seton Healthcare Family (Other); Texas Department of State Health Services (Other); Duke University (Other); City University of New York, School of Public Health (Other)
Responsible Party: Principal Investigator, Deanna Hoelscher, John P McGovern Professor in Health Promotion and Director, Michael & Susan Dell Center for Healthy Living, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-SPH-11-0513 RCT
Record Dates: First submitted 2016-03-08; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Childhood Obesity
Keywords: child obesity; primary prevention; primary care; weight management; child overweight; BMI
MeSH Terms: conditions — Pediatric Obesity | interventions — Body Mass Index; Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TX CORD Intervention (Experimental): TX CORD Intervention. The intervention entailed: (1) BMI screening, (2) Next Steps brief counseling materials for the healthcare provider, (3) a 3-month intensive Mind Exercise Nutrition Do It! and Coordinated Approach To Child Health (MEND/CATCH) phase, which included the Mind Exercise Nutrition Do it! ( MEND) programs for preschool (ages 2-5) and school-aged (ages 6-12) children coupled with adapted CATCH activities, and (5) a 9-month transition MEND/CATCH Transition phase, which offered monthly reinforcement sessions for parents and children, and twice weekly Young Men's Christian Association (YMCA) sports for children. Community Health Workers (CHWs) serve as program liaisons and assist in delivering all intervention group sessions as well as tracking families. Electronic Health Record (EHR) changes supported the screening and Next Steps delivery.
  Interventions: Behavioral: BMI screening; Behavioral: Next Steps brief clinical intervention; Behavioral: MEND/CATCH; Behavioral: MEND/CATCH Transition Phase
- Brief Clinic Comparison (Active Comparator): Next Steps brief clinical intervention. The comparison program was a 12-month clinic-based program conducted at twelve partner healthcare clinics and entailed (1) EHR changes to support childhood obesity clinical visits; (2) BMI screening, (3) Next Steps brief counseling materials for the healthcare provider, and (4) Next Steps self-paced booklet for parents and children to work on nutrition and physical activity targets in a self-directed manner. Families were encouraged to seek repeated clinical visits to address child obesity.
  Interventions: Behavioral: BMI screening; Behavioral: Next Steps brief clinical intervention; Behavioral: Next Steps Self-Paced Booklet

INTERVENTIONS:
Behavioral: BMI screening — Physician screening of patients to identify patients who are overweight or obese.
  Other Names: Body Mass Index (BMI) Screening
Behavioral: Next Steps brief clinical intervention — This intervention included identification of children who were overweight or obese, and Next Steps brief counseling materials for the healthcare provider (prior to enrollment in the intervention).
  Other Names: Next Steps
Behavioral: MEND/CATCH — MEND 2-5 and MEND/CATCH 6-12 programs are multi-component interventions including behavioral, nutrition, and physical activity sessions. In the intensive (first 3 months) phase, MEND 2-5 entailed nine weekly sessions and MEND 6-12 entailed 18 twice weekly sessions.
  Other Names: Mind Exercise Nutrition Do it! (MEND); Coordinated Approach To Child Health (CATCH)
  Arms: TX CORD Intervention
Behavioral: MEND/CATCH Transition Phase — The transition phase (next 9 months of the 12-month program) included monthly 90-minute sessions for parents and children included MEND reviews, cooking classes, Being Well book, CATCH activities and MEND World activities. Children were enrolled in YMCA sports teams or programs offered twice weekly to encourage physical activity. Weekly text messages were sent to parents to reinforce behavioral objectives of the intervention.
  Arms: TX CORD Intervention
Behavioral: Next Steps Self-Paced Booklet — Next Steps booklet for parents and children to work on nutrition and physical activity targets in a self-directed manner. Families were encouraged to seek repeated clinical visits to address child obesity as a follow up to the self-paced booklet.
  Other Names: Next Steps Workbook
  Arms: Brief Clinic Comparison

SUMMARY:
A systems approach emphasizes the linkage between individual behavior change strategies and social and physical environmental changes, which act synergistically to facilitate (or inhibit) healthy eating and active living. The hypothesis of this study is that among low-income, ethnically diverse overweight and obese children, aged 2-12 years, a systems approach to child obesity will reduce body mass index (BMI) compared to primary prevention alone.

DETAILED DESCRIPTION:
The goal of this project is to develop, implement and evaluate an integrated, systems-oriented obesity model for underserved, ethnically diverse children aged 2-12 years. The first step will include conducting an assets-based community assessment in low-income neighborhood catchment areas in Austin and Houston, TX with input and data-sharing from existing partnerships. Results from this assessment will inform and facilitate the implementation of both primary and secondary prevention efforts across multiple sectors (healthcare, school, and childcare). The demonstration project will include secondary prevention programs embedded within community primary prevention efforts. For primary prevention, a quasi-experimental approach will be used, where existing obesity prevention efforts are reinforced and optimized in healthcare clinics, Head Start Centers and schools in the catchment areas (NOTE: the primary prevention intervention study is further described in ClinicalTrials.gov at Texas Childhood Obesity Research Demonstration project Primary Prevention Intervention {TXCORDPRIM) under a different protocol & record). Secondary prevention includes integration of the investigative team's evidence-based portfolio of family and community interventions, specifically the MEND/CATCH programs. For secondary prevention, a randomized controlled trial design will be used in which individual overweight/obese children are randomized to a 12-month community-centered, family-based obesity program or to primary prevention alone.

The hypothesis of this study is that among low-income, ethnically diverse overweight and obese children, aged 2-12 years, a systems approach to child obesity will reduce body mass index (BMI, expressed as %95th percentile) compared to primary prevention alone. The specific aims of the grant are as follows (see below).

Aim 1: To implement and evaluate the efficacy of a systems approach to child obesity on reducing BMI (expressed as %95th percentile) by embedding a 12-month family-based secondary prevention program within a community primary prevention program. The secondary prevention weight management program will target overweight/obese children and their families in the primary prevention catchment areas in Austin and Houston. Overweight/obese children (total n=576), aged 2-12 years, will be randomly assigned to either the 12-month secondary prevention program (experimental) or the community primary prevention program alone (control), in equal age subgroups (2-5, 6-8, and 9-12 years). Analyses will be conducted by age group, and outcomes will include BMI as expressed as %95th percentile), obesity-related behaviors, quality of life, and program use indicators.

Aim 2: To quantify the incremental cost-effectiveness of the 12-month family-based secondary prevention program relative to primary prevention alone for child obesity. Activity Based Costing methods will be used to quantify the incremental cost of delivering the secondary prevention program relative to optimized healthcare. These costs will then be combined with the effectiveness data to quantify the incremental cost-effectiveness of the community-based intervention.

All project activities will be coordinated with input from Demonstration Project Research Network Committee (CDC and the Evaluation Center).

ELIGIBILITY:
Inclusion Criteria:

* 2-12 years of age and
* ≥ 85th percentile for BMI

Exclusion Criteria:

* complications of obesity that would interfere with participation (e.g., severe respiratory insufficiency or orthopedic problems);
* underlying obesity-related conditions, such as systemic steroid use or endocrine abnormalities;
* severe psychological problems; and
* participation in an obesity treatment program within the past year.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 549 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in obesity as indicated by body mass index (BMI) expressed as %95th percentile | Baseline to 3 months
  Body mass index (BMI), expressed as %95th BMI percentile
Change in obesity as indicated by body mass index (BMI) expressed as %95th percentile | 3 months to 12 months
  Body mass index (BMI), expressed as %95th BMI percentile

OTHER OUTCOMES:
Change in Waist:height ratio | Baseline to 3 months
  Waist:height (ratio), each measured in cm
Change in Waist:height ratio | 3 months to 12 months
  Waist:height (ratio), each measured in cm
Change in Fat free mass in kg | Baseline to 3 months
  Fat free mass (kg) is defined as total body weight minus weight of body fat
Change in Fat free mass in kg | 3 months to 12 months
  Fat free mass (kg) is defined as total body weight minus weight of body fat
Change in Fat mass in kg and percent | Baseline to 3 months
  Fat mass (kg and %) is the body weight of fat
Change in Fat mass in kg and percent | 3 months to 12 months
  Fat mass (kg and %) is the body weight of fat
Change in Systolic blood pressure | Baseline to 3 months
  Systolic blood pressure (mmHg)
Change in Systolic blood pressure | 3 months to 12 months
  Systolic blood pressure (mmHg)
Change in Diastolic blood pressure | Baseline to 3 months
  Diastolic blood pressure (mmHg)
Change in Diastolic blood pressure | 3 months to 12 months
  Diastolic blood pressure (mmHg)
Change in Fitness as indicated by heart rate (post exercise 1 minute) | Baseline to 3 months
  Heart rate (post step test exercise 1 min)
Change in Fitness as indicated by heart rate (post exercise 1 minute) | 3 months to 12 months
  Heart rate (post step test exercise 1 min)
Change in Quality of Life as assessed by the Child Quality of Life (QOL) scale | Baseline to 3 months
  Child Quality of Life (QOL) scale
Change in Quality of Life as assessed by the Child Quality of Life (QOL) scale | 3 months to 12 months
  Child Quality of Life (QOL) scale

CONTACTS AND LOCATIONS:
Overall Officials: Deanna M Hoelscher, PhD, Principal Investigator — The University of Texas Health Science Center, Houston; Nancy F Butte, PhD, Principal Investigator — Children's Nutrition Research Center, Baylor College of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoelscher DM, Butte NF, Barlow S, Vandewater EA, Sharma SV, Huang T, Finkelstein E, Pont S, Sacher P, Byrd-Williams C, Oluyomi AO, Durand C, Li L, Kelder SH. Incorporating primary and secondary prevention approaches to address childhood obesity prevention and treatment in a low-income, ethnically diverse population: study design and demographic data from the Texas Childhood Obesity Research Demonstration (TX CORD) study. Child Obes. 2015 Feb;11(1):71-91. doi: 10.1089/chi.2014.0084. Epub 2015 Jan 2. PMID 25555188
- [Background] Oluyomi AO, Byars A, Byrd-Williams C, Sharma SV, Durand C, Hoelscher DM, Butte NF, Kelder SH. The utility of Geographical Information Systems (GIS) in systems-oriented obesity intervention projects: the selection of comparable study sites for a quasi-experimental intervention design--TX CORD. Child Obes. 2015 Feb;11(1):58-70. doi: 10.1089/chi.2014.0054. Epub 2015 Jan 14. PMID 25587670
- [Derived] Barlow SE, Salahuddin M, Durand C, Pont SJ, Hoelscher DM, Butte NF. Evaluation of BMI Metrics to Assess Change in Adiposity in Children with Overweight and Moderate and Severe Obesity. Obesity (Silver Spring). 2020 Aug;28(8):1512-1518. doi: 10.1002/oby.22858. Epub 2020 Jul 6. PMID 32935936
- [Derived] Barlow SE, Durand C, Salahuddin M, Pont SJ, Butte NF, Hoelscher DM. Who benefits from the intervention? Correlates of successful BMI reduction in the Texas Childhood Obesity Demonstration Project (TX-CORD). Pediatr Obes. 2020 May;15(5):e12609. doi: 10.1111/ijpo.12609. Epub 2020 Jan 15. PMID 31944617
- [Derived] Butte NF, Hoelscher DM, Barlow SE, Pont S, Durand C, Vandewater EA, Liu Y, Adolph AL, Perez A, Wilson TA, Gonzalez A, Puyau MR, Sharma SV, Byrd-Williams C, Oluyomi A, Huang T, Finkelstein EA, Sacher PM, Kelder SH. Efficacy of a Community- Versus Primary Care-Centered Program for Childhood Obesity: TX CORD RCT. Obesity (Silver Spring). 2017 Sep;25(9):1584-1593. doi: 10.1002/oby.21929. Epub 2017 Jul 13. PMID 28703504